CLINICAL TRIAL: NCT07386548
Title: Bone Marrow Aspirate Concentrate Injection With MRI's - A Prospective Randomized Control Trial
Brief Title: Biologic Injection For Adults With Lumbar Disc Herniation
Acronym: BMAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Aclarion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-09027977
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Degenerative Disc Disease; DDD; Degenerative Disc Disease Lumbar; Degenerative Disc Disease, Lumbar; Lumbar Disc Herniation; Disc Herniation, Lumbar; Bone Marrow Aspirate Concentrate; Intervertebral Disc Displacement; Low Back Pain; Chronic Low Back Pain (CLBP); CLBP - Chronic Low Back Pain
Keywords: degenerative disc disease; lumbar disc herniation; bone marrow aspirate concentrate; intervertebral disc displacement; low back pain
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral Disc Displacement; Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMAC Group (Active Comparator): Administration of one 1-2cc intradiscal Bone Marrow Aspirate Concentrate (BMAC) injection during lumbar microdiscectomy surgery.
  Interventions: Other: Bone Marrow Aspirate Concentrate (BMAC)
- Control Group (No Intervention): Standard of care lumbar microdiscectomy surgery without the BMAC injection.

INTERVENTIONS:
Other: Bone Marrow Aspirate Concentrate (BMAC) — Dosage Form: Autologous intradiscal injection Dosage: 1-2 cc's Frequency: Once, during surgery Duration: N/A
  Other Names: Bone Marrow Aspirate (BMA); Bone Marrow Aspirate Stem Cell Concentrate (BMAC); Bone Marrow Concentrate (BMC)
  Arms: BMAC Group

SUMMARY:
The goal of this clinical trial is to find out whether adding a bone-marrow aspirate concentrate (BMAC) injection during surgery can improve recovery in adults undergoing lumbar microdiscectomy for a lumbar disc herniation.

The main questions it aims to answer are:

* Does the BMAC injection lead to better disc tissue health after surgery (as seen on MRI scans)?
* Does the BMAC injection lead to greater improvement in pain and disability compared to surgery alone?

Participants will be adults aged 18 and older who are scheduled for lumbar microdiscectomy surgery.

Researchers will compare one group of participants receiving the standard-of-care surgery plus the BMAC injection with another group receiving the same surgery without the injection to see if the injection offers added benefit.

Participants will:

* Have surgery (microdiscectomy) with or without the injection.
* Complete pain and disability questionnaires at several times over 2 years.
* Undergo MRI scans at baseline and follow-up to assess disc structure and tissue health.
* Provide samples of leftover disc or bone-marrow tissue (as applicable) from surgery for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* Clinically and/or radiographically (MRI) confirmed diagnosis of degenerative disc disease of the lumbar spine, lumbar disc herniation, and indication for lumbar microdiscectomy surgery
* Unresponsive to conservative/non-operative treatment for >3 months
* Psychosocial, mental and physical ability to understand and to adhere to this protocol, especially adhering to the visit schedule follow-ups and observe the treatment plan

Exclusion Criteria:

* Prisoners
* Individuals who are not yet adults (infants, children, teenagers)
* Individuals who are not able to clearly understand English
* Adults with diminished capacity to consent
* Major cognitive impairment causing to inability to understand and provide informed consent
* Active malignancy
* Active chronic or acute infection
* Autoimmune disorder that impacts the lumbar spine (ankylosing spondylitis, lupus e.g.)
* Bone marrow-derived or non-bone marrow-derived cancer
* Low platelet count or clotting disorders
* Prior surgery at the level to be treated or the adjacent level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Intervertebral Disc Hydration at 3 Months | Baseline and 3 Months post-operation
  MRI T2 mapping and T2 relaxation time are advanced imaging techniques that help assess the hydration status of intervertebral discs. These two metrics will be combined as one data point. T2 relaxation time measures the decay of the MRI signal, which is influenced by the water content in the disc. Higher T2 values indicate better hydration, while lower T2 values suggest dehydration and degeneration. T2 mapping provides a detailed, quantitative assessment of the disc's water content, allowing for early detection of degenerative changes before they become visible on standard MRI images. This information is crucial for diagnosing the extent of disc degeneration, planning surgical interventions, and monitoring the effectiveness of treatments aimed at restoring disc health.
Change from Baseline in Intervertebral Disc Hydration at 1 Year | Baseline and 1 year post-operation
  MRI T2 mapping and T2 relaxation time are advanced imaging techniques that help assess the hydration status of intervertebral discs. These two metrics will be combined as one data point. T2 relaxation time measures the decay of the MRI signal, which is influenced by the water content in the disc. Higher T2 values indicate better hydration, while lower T2 values suggest dehydration and degeneration. T2 mapping provides a detailed, quantitative assessment of the disc's water content, allowing for early detection of degenerative changes before they become visible on standard MRI images. This information is crucial for diagnosing the extent of disc degeneration, planning surgical interventions, and monitoring the effectiveness of treatments aimed at restoring disc health.
Change from Baseline in Intervertebral Disc Hydration at 2 Years | Baseline and 2 years post-operation
  MRI T2 mapping and T2 relaxation time are advanced imaging techniques that help assess the hydration status of intervertebral discs. These two metrics will be combined as one data point. T2 relaxation time measures the decay of the MRI signal, which is influenced by the water content in the disc. Higher T2 values indicate better hydration, while lower T2 values suggest dehydration and degeneration. T2 mapping provides a detailed, quantitative assessment of the disc's water content, allowing for early detection of degenerative changes before they become visible on standard MRI images. This information is crucial for diagnosing the extent of disc degeneration, planning surgical interventions, and monitoring the effectiveness of treatments aimed at restoring disc health.
Change from Baseline in Proteoglycan Content at 3 Months | From enrollment to 3 Months post-operation
  MRI T1 rho mapping and T1 rho relaxation time are advanced imaging techniques that provide insights into the biochemical composition of intervertebral discs, particularly the proteoglycan content. T1 rho relaxation time measures the decay of the MRI signal in the presence of a spin-lock pulse, which is sensitive to interactions between water molecules and macromolecules like proteoglycans. These two metrics will be combined as one data point. Higher T1 rho values indicate higher proteoglycan content and better disc hydration, while lower values suggest degeneration and reduced proteoglycan levels. T1 rho mapping offers a detailed, quantitative assessment of these biochemical changes, allowing for early detection of disc degeneration and aiding in the evaluation of treatment efficacy.
Change from Baseline in Proteoglycan Content at 1 Year | From enrollment to 1 year post-operation
  MRI T1 rho mapping and T1 rho relaxation time are advanced imaging techniques that provide insights into the biochemical composition of intervertebral discs, particularly the proteoglycan content. T1 rho relaxation time measures the decay of the MRI signal in the presence of a spin-lock pulse, which is sensitive to interactions between water molecules and macromolecules like proteoglycans. These two metrics will be combined as one data point. Higher T1 rho values indicate higher proteoglycan content and better disc hydration, while lower values suggest degeneration and reduced proteoglycan levels. T1 rho mapping offers a detailed, quantitative assessment of these biochemical changes, allowing for early detection of disc degeneration and aiding in the evaluation of treatment efficacy.
Change from Baseline in Proteoglycan Content at 2 Years | From enrollment to 2 years post-operation
  MRI T1 rho mapping and T1 rho relaxation time are advanced imaging techniques that provide insights into the biochemical composition of intervertebral discs, particularly the proteoglycan content. T1 rho relaxation time measures the decay of the MRI signal in the presence of a spin-lock pulse, which is sensitive to interactions between water molecules and macromolecules like proteoglycans. These two metrics will be combined as one data point. Higher T1 rho values indicate higher proteoglycan content and better disc hydration, while lower values suggest degeneration and reduced proteoglycan levels. T1 rho mapping offers a detailed, quantitative assessment of these biochemical changes, allowing for early detection of disc degeneration and aiding in the evaluation of treatment efficacy.
Change from Baseline in Disc Height Index at 3 Months | From enrollment to 3 months post-operation
  Assessed via MRI, the Disc Height Index (DHI) is a measurement used in spine surgery to assess the height of an intervertebral disc. It is calculated by dividing the height of the disc at the mid-vertebral line by the height of the superior vertebral body. This index helps in evaluating the degree of disc degeneration and is often used to monitor changes before and after surgical interventions.
Change from Baseline in Disc Height Index at 1 Year | From enrollment to 1 year post-operation
  Assessed via MRI, the Disc Height Index (DHI) is a measurement used in spine surgery to assess the height of an intervertebral disc. It is calculated by dividing the height of the disc at the mid-vertebral line by the height of the superior vertebral body. This index helps in evaluating the degree of disc degeneration and is often used to monitor changes before and after surgical interventions.
Change from Baseline in Disc Height Index at 2 Years | From enrollment to 2 years post-operation
  Assessed via MRI, the Disc Height Index (DHI) is a measurement used in spine surgery to assess the height of an intervertebral disc. It is calculated by dividing the height of the disc at the mid-vertebral line by the height of the superior vertebral body. This index helps in evaluating the degree of disc degeneration and is often used to monitor changes before and after surgical interventions.
Change from Baseline in Pfirrmann Grade at 3 Months | From enrollment to 3 months post-operation
  Assessed via MRI, Pfirrmann grading is a radiological classification used to assess the severity of lumbar intervertebral disc degeneration. It categorizes disc degeneration into five grades based on specific criteria related to the appearance of the discs:
  Grade I: Normal disc with high signal intensity and well-defined nucleus and annulus.
  Grade II: Slightly degenerated disc with a normal height but a lower signal intensity in the nucleus.
  Grade III: Moderate degeneration with a loss of disc height and a more pronounced decrease in signal intensity.
  Grade IV: Severe degeneration with significant loss of disc height and a very low signal intensity.
  Grade V: End-stage degeneration with a collapsed disc and no visible nucleus
Change from Baseline in Pfirrmann Grade at 1 Year | From enrollment to 1 year post-operation
  Assessed via MRI, Pfirrmann grading is a radiological classification used to assess the severity of lumbar intervertebral disc degeneration. It categorizes disc degeneration into five grades based on specific criteria related to the appearance of the discs:
  Grade I: Normal disc with high signal intensity and well-defined nucleus and annulus.
  Grade II: Slightly degenerated disc with a normal height but a lower signal intensity in the nucleus.
  Grade III: Moderate degeneration with a loss of disc height and a more pronounced decrease in signal intensity.
  Grade IV: Severe degeneration with significant loss of disc height and a very low signal intensity.
  Grade V: End-stage degeneration with a collapsed disc and no visible nucleus
Change from Baseline in Pfirrmann Grade at 2 Years | From enrollment to 2 years post-operation
  Assessed via MRI, Pfirrmann grading is a radiological classification used to assess the severity of lumbar intervertebral disc degeneration. It categorizes disc degeneration into five grades based on specific criteria related to the appearance of the discs:
  Grade I: Normal disc with high signal intensity and well-defined nucleus and annulus.
  Grade II: Slightly degenerated disc with a normal height but a lower signal intensity in the nucleus.
  Grade III: Moderate degeneration with a loss of disc height and a more pronounced decrease in signal intensity.
  Grade IV: Severe degeneration with significant loss of disc height and a very low signal intensity.
  Grade V: End-stage degeneration with a collapsed disc and no visible nucleus
Change from Baseline in Nucleus Pulposus Size at 3 Months | From enrollment to 3 months post-operation
  The Nucleus Pulposus is the soft, gel-like center of an intervertebral disc, surrounded by the tougher annulus fibrosus. It plays a crucial role in absorbing shock and allowing flexibility in the spine. Assessed via MRI, the size and condition of the nucleus pulposus are indicators of disc health. A healthy nucleus pulposus is typically well-hydrated and maintains disc height, while a degenerated nucleus pulposus may shrink and lose its cushioning ability.
Change from Baseline in Nucleus Pulposus Size at 1 Year | From enrollment to 1 year post-operation
  The Nucleus Pulposus is the soft, gel-like center of an intervertebral disc, surrounded by the tougher annulus fibrosus. It plays a crucial role in absorbing shock and allowing flexibility in the spine. Assessed via MRI, the size and condition of the nucleus pulposus are indicators of disc health. A healthy nucleus pulposus is typically well-hydrated and maintains disc height, while a degenerated nucleus pulposus may shrink and lose its cushioning ability.
Change from Baseline in Nucleus Pulposus Size at 2 Years | From enrollment to 2 years post-operation
  The Nucleus Pulposus is the soft, gel-like center of an intervertebral disc, surrounded by the tougher annulus fibrosus. It plays a crucial role in absorbing shock and allowing flexibility in the spine. Assessed via MRI, the size and condition of the nucleus pulposus are indicators of disc health. A healthy nucleus pulposus is typically well-hydrated and maintains disc height, while a degenerated nucleus pulposus may shrink and lose its cushioning ability.
Change from Baseline in NOCISCORE at 3 Months | From enrollment to 3 months post-operation
  Assessed via MRI, decreases in pain biomarkers within the intervertebral disc will be measured using Magnetic Resonance Spectroscopy (MRS). MRS is non-invasive. The data is analyzed and summarized in a NOCIGRAM report, which provides an objective analysis of the pain biomarkers observed during a preoperative MRI scan.
  The NOCISCORE measures six biomarker ratios associated with pain generation for each disc. The scores for each disc level are categorized into NOCI+, Mild, and NOCI-, from most 'painful' to 'least painful' levels.
Change from Baseline in NOCISCORE at 1 Year | From enrollment to 1 year post-operation
  Assessed via MRI, decreases in pain biomarkers within the intervertebral disc will be measured using Magnetic Resonance Spectroscopy (MRS). MRS is non-invasive. The data is analyzed and summarized in a NOCIGRAM report, which provides an objective analysis of the pain biomarkers observed during a preoperative MRI scan.
  The NOCISCORE measures six biomarker ratios associated with pain generation for each disc. The scores for each disc level are categorized into NOCI+, Mild, and NOCI-, from most 'painful' to 'least painful' levels.
Change from Baseline in NOCISCORE at 2 Years | From enrollment to 2 years post-operation
  Assessed via MRI, decreases in pain biomarkers within the intervertebral disc will be measured using Magnetic Resonance Spectroscopy (MRS). MRS is non-invasive. The data is analyzed and summarized in a NOCIGRAM report, which provides an objective analysis of the pain biomarkers observed during a preoperative MRI scan.
  The NOCISCORE measures six biomarker ratios associated with pain generation for each disc. The scores for each disc level are categorized into NOCI+, Mild, and NOCI-, from most 'painful' to 'least painful' levels.

SECONDARY OUTCOMES:
Change from Baseline in Patient Reported Pain at 3 Months | From enrollment to 3 Months post-operation
  The Numeric Rating Scale (NRS) is one of the most commonly used pain scales in medicine. It can be administered verbally or self-administered on paper. Zero is equivalent to no pain and 10 indicates the worst possible pain.
Change from Baseline in Patient Reported Pain at 6 Months | From enrollment to 6 Months post-operation
  The Numeric Rating Scale (NRS) is one of the most commonly used pain scales in medicine. It can be administered verbally or self-administered on paper. Zero is equivalent to no pain and 10 indicates the worst possible pain.
Change from Baseline in Patient Reported Pain at 1 Year | From enrollment to 1 Year post-operation
  The Numeric Rating Scale (NRS) is one of the most commonly used pain scales in medicine. It can be administered verbally or self-administered on paper. Zero is equivalent to no pain and 10 indicates the worst possible pain.
Change from Baseline in Patient Reported Pain at 2 Years | From enrollment to 2 years post-operation
  The Numeric Rating Scale (NRS) is one of the most commonly used pain scales in medicine. It can be administered verbally or self-administered on paper. Zero is equivalent to no pain and 10 indicates the worst possible pain.
Change from Baseline in Patient Reported Disability at 3 Months | From enrollment to 3 Months post-operation
  The Oswestry Disability Index (ODI) is a self-administered questionnaire divided into ten sections designed to assess limitations in various aspects of daily living activities. Each section is scored from 0 to 5, where 0 indicates no disability and 5 indicates maximum disability. The total score is calculated as a percentage ranging from 0% (no disability) to 100% (maximum disability).
Change from Baseline in Patient Reported Disability at 6 Months | From enrollment to 6 Months post-operation
  The Oswestry Disability Index (ODI) is a self-administered questionnaire divided into ten sections designed to assess limitations in various aspects of daily living activities. Each section is scored from 0 to 5, where 0 indicates no disability and 5 indicates maximum disability. The total score is calculated as a percentage ranging from 0% (no disability) to 100% (maximum disability).
Change from Baseline in Patient Reported Disability at 1 Year | From enrollment to 1 year post-operation
  The Oswestry Disability Index (ODI) is a self-administered questionnaire divided into ten sections designed to assess limitations in various aspects of daily living activities. Each section is scored from 0 to 5, where 0 indicates no disability and 5 indicates maximum disability. The total score is calculated as a percentage ranging from 0% (no disability) to 100% (maximum disability).
Change from Baseline in Patient Reported Disability at 2 Years | From enrollment to 2 years post-operation
  The Oswestry Disability Index (ODI) is a self-administered questionnaire divided into ten sections designed to assess limitations in various aspects of daily living activities. Each section is scored from 0 to 5, where 0 indicates no disability and 5 indicates maximum disability. The total score is calculated as a percentage ranging from 0% (no disability) to 100% (maximum disability).
Change from Baseline in SI-Score at 3 Months | From enrollment to 3 months post-operation
  Assessed via MRI, decreases in pain biomarkers within the intervertebral disc will be measured using Magnetic Resonance Spectroscopy (MRS). MRS is non-invasive. The data is analyzed and summarized in a NOCIGRAM report, which provides an objective analysis of the pain biomarkers observed during a preoperative MRI scan.
  The SI-Score (Structural Integrity Score) reflects the relative amounts of proteoglycan between discs as an indication of relative structural integrity between the discs on a scale from 0 to 1. Higher SI scores reflect higher relative values as compared between discs in the patient and do not necessarily reflect high structural integrity. A low SI score, corresponding to a lower structural integrity, is associated with more advanced degeneration (relative between discs).
Change from Baseline in SI-Score at 1 Year | From enrollment to 1 year post-operation
  Assessed via MRI, decreases in pain biomarkers within the intervertebral disc will be measured using Magnetic Resonance Spectroscopy (MRS). MRS is non-invasive. The data is analyzed and summarized in a NOCIGRAM report, which provides an objective analysis of the pain biomarkers observed during a preoperative MRI scan.
  The SI-Score (Structural Integrity Score) reflects the relative amounts of proteoglycan between discs as an indication of relative structural integrity between the discs on a scale from 0 to 1. Higher SI scores reflect higher relative values as compared between discs in the patient and do not necessarily reflect high structural integrity. A low SI score, corresponding to a lower structural integrity, is associated with more advanced degeneration (relative between discs).
Change from Baseline in SI-Score at 2 Years | From enrollment to 2 years post-operation
  Assessed via MRI, decreases in pain biomarkers within the intervertebral disc will be measured using Magnetic Resonance Spectroscopy (MRS). MRS is non-invasive. The data is analyzed and summarized in a NOCIGRAM report, which provides an objective analysis of the pain biomarkers observed during a preoperative MRI scan.
  The SI-Score (Structural Integrity Score) reflects the relative amounts of proteoglycan between discs as an indication of relative structural integrity between the discs on a scale from 0 to 1. Higher SI scores reflect higher relative values as compared between discs in the patient and do not necessarily reflect high structural integrity. A low SI score, corresponding to a lower structural integrity, is associated with more advanced degeneration (relative between discs).

CONTACTS AND LOCATIONS:
Overall Officials: Roger Hartl, MD, Principal Investigator — NewYork Presbyterian-Weill Cornell Medicine
Locations (1):
- NewYork-Presbyterian/Weill Cornell Medical Center, Manhattan, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data, for any purpose, may do so indefinitely at (Link to be included).

REFERENCES:
- [Background] Zhang W, Sun T, Li Y, Yang M, Zhao Y, Liu J, Li Z. Application of stem cells in the repair of intervertebral disc degeneration. Stem Cell Res Ther. 2022 Feb 11;13(1):70. doi: 10.1186/s13287-022-02745-y. PMID 35148808
- [Background] Elabd C, Centeno CJ, Schultz JR, Lutz G, Ichim T, Silva FJ. Intra-discal injection of autologous, hypoxic cultured bone marrow-derived mesenchymal stem cells in five patients with chronic lower back pain: a long-term safety and feasibility study. J Transl Med. 2016 Sep 1;14(1):253. doi: 10.1186/s12967-016-1015-5. PMID 27585696
- [Background] Mochida J, Sakai D, Nakamura Y, Watanabe T, Yamamoto Y, Kato S. Intervertebral disc repair with activated nucleus pulposus cell transplantation: a three-year, prospective clinical study of its safety. Eur Cell Mater. 2015 Mar 20;29:202-12; discussion 212. doi: 10.22203/ecm.v029a15. PMID 25794529
- [Background] Noriega DC, Ardura F, Hernandez-Ramajo R, Martin-Ferrero MA, Sanchez-Lite I, Toribio B, Alberca M, Garcia V, Moraleda JM, Gonzalez-Vallinas M, Sanchez A, Garcia-Sancho J. Treatment of Degenerative Disc Disease With Allogeneic Mesenchymal Stem Cells: Long-term Follow-up Results. Transplantation. 2021 Feb 1;105(2):e25-e27. doi: 10.1097/TP.0000000000003471. No abstract available. PMID 33492116
- [Background] Jerome MA, Lutz C, Lutz GE. Risks of Intradiscal Orthobiologic Injections: A Review of the Literature and Case Series Presentation. Int J Spine Surg. 2021 Apr;15(s1):26-39. doi: 10.14444/8053. Epub 2021 Apr 21. PMID 34376494
- [Background] Pettine KA, Murphy MB, Suzuki RK, Sand TT. Percutaneous injection of autologous bone marrow concentrate cells significantly reduces lumbar discogenic pain through 12 months. Stem Cells. 2015 Jan;33(1):146-56. doi: 10.1002/stem.1845. PMID 25187512
- [Background] Yoshikawa T, Ueda Y, Miyazaki K, Koizumi M, Takakura Y. Disc regeneration therapy using marrow mesenchymal cell transplantation: a report of two case studies. Spine (Phila Pa 1976). 2010 May 15;35(11):E475-80. doi: 10.1097/BRS.0b013e3181cd2cf4. PMID 20421856
- [Background] Orozco L, Soler R, Morera C, Alberca M, Sanchez A, Garcia-Sancho J. Intervertebral disc repair by autologous mesenchymal bone marrow cells: a pilot study. Transplantation. 2011 Oct 15;92(7):822-8. doi: 10.1097/TP.0b013e3182298a15. PMID 21792091
- [Background] Comella K, Silbert R, Parlo M. Effects of the intradiscal implantation of stromal vascular fraction plus platelet rich plasma in patients with degenerative disc disease. J Transl Med. 2017 Jan 13;15(1):12. doi: 10.1186/s12967-016-1109-0. PMID 28086781
- See also: Cleveland Clinic: Bone Marrow Concentrate (BMC) — https://my.clevelandclinic.org/health/procedures/bone-marrow-concentrate-bmc